CLINICAL TRIAL: NCT00416182
Title: The Use of Nasally Delivered Pulmozyme in the Treatment of Sinusitis in Cystic Fibrosis Patients: A Pilot Study
Brief Title: Nasally Delivered Pulmozyme for Sinusitis in Cystic Fibrosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Vermont (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Thomas Lahiri, Professor of Pediatrics, University of Vermont
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Z3297S
Record Dates: First submitted 2006-12-26; First posted 2006-12-27 (Estimated); Results first posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Sinusitis; Cystic Fibrosis
Keywords: Cystic fibrosis; chronic sinusitis; mucolytic
MeSH Terms: conditions — Sinusitis; Cystic Fibrosis | interventions — dornase alfa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pulmozyme (Experimental): 2.5 mg Pulmozyme (dornase alfa) delivered intranasally once daily
  Interventions: Drug: Pulmozyme (dornase alfa)
- placebo (Placebo Comparator): 2.5 mg/2mL placebo administered intranasally once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pulmozyme (dornase alfa) — 2.5 mg/2.5 mL of Pulmozyme (dornase alfa) delivered via Sinustar nasal nebulizer device
  Other Names: Pulmozyme, dornase alfa, human recombinant DNase 1
  Arms: Pulmozyme
Drug: Placebo — 2.5 mL of placebo delivered via Sinustar nebulizer device
  Other Names: placebo comparator
  Arms: placebo

SUMMARY:
Chronic sinusitis is a frequent complication in cystic fibrosis. The aim of this study is to determine whether Pulmozyme(dornase alfa) would maintain sinus health (compared to placebo) in patients with cystic fibrosis who have recently undergone sinus surgery.

DETAILED DESCRIPTION:
AIM: To evaluate the effectiveness of Pulmozyme(dornase alfa) in decreasing post-operative sinusitis symptoms in patients with cystic fibrosis (CF)

PROCEDURES: 20 patients with CF will be randomized to receive either Pulmozyme or placebo via nasal inhalation daily for 12 months. Consent will be obtained following surgery and treatment will begin 1 week post-operatively.

Monitoring will include examination and recording of adverse effects and follow up weekly for one month and then at 2.5, 6, 9 and 12 months.

Outcome measures will include ciliary function testing, pulmonary function testing, sinus questionnaires and CT scan.

ELIGIBILITY:
Inclusion Criteria:

* Clinical and laboratory diagnosis of cystic fibrosis
* Age greater than or equal to 5 years
* Forced expiratory volume in 1 second (FEV1) greater than or equal to 40% predicted
* Sinus surgery within one week of enrollment

Exclusion Criteria:

* Pregnancy
* Intolerance of orally inhaled Pulmozyme (dornase alfa)

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2006-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Lahiri, MD, Principal Investigator — University of Vermont; Sandra Diehl, MS, Study Director — University of Vermont Medical Center
Locations (1):
- Fletcher Allen Health Care, Burlington, Vermont, United States

REFERENCES:
- [Result] Lahiri T, Herrington H, Diehl S, Landrigan G. The effect of intranasal dornase alfa on chronic sinusitis in patients with cystic fibrosis: a pilot study. Pediatr Pulmonol S35:354, 2012.
- [Derived] Yang C, Montgomery M. Dornase alfa for cystic fibrosis. Cochrane Database Syst Rev. 2021 Mar 18;3(3):CD001127. doi: 10.1002/14651858.CD001127.pub5. PMID 33735508

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients undergoing sinus surgery meeting inclusion criteria were approached in the outpatient or hospital setting
Pre-assignment Details: upon providing informed consent, subjects were randomized and blinded to treatment or placebo groups
Groups:
- Pulmozyme (Dornase Alfa): 2.5 mg/2.5mL of Pulmozyme administered intranasally once daily
- Placebo: 2.5mg/2.5mL placebo administered intranasally once daily
Period: Overall Study
Arm/Group | Pulmozyme (Dornase Alfa) | Placebo
Started | 8 | 8
Completed | 5 | 6
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Pulmozyme (Dornase Alfa): 2.5 mg/2.5 mL of intranasal Pulmozyme
- Placebo: 2.5 mL of placebo comparator
- Total: Total of all reporting groups
Arm/Group | Pulmozyme (Dornase Alfa) | Placebo | Total
Number analyzed (Participants) | 8 | 8 | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 6 | 9
  Between 18 and 65 years | 5 | 2 | 7
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 5 | 10
  Male | 3 | 3 | 6
Region of Enrollment [Number; unit: participants]
  United States | 8 | 8 | 16

OUTCOME MEASURES:

1. Primary Outcome: Computed Tomography Evidence of Less Sinus Disease
Description: compare sinus CT pre-op (baseline) to one year after initiation of study drug Difference in pre and post scores by Lund-McKay scoring system are reported (1 year minus baseline) The Lund-Mackay scoring system was used to evaluate the extent and severity of sinusitis. The scale ranges from 0 (best possible outcome with complete lucency of all sinuses) to 24 (worst possible outcome with complete opacification of all sinuses)
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Pulmozyme: Patients receiving 2.5 mg intranasal Pulmozyme once daily
- Placebo: Patients receiving intranasal placebo once daily
Arm/Group | Pulmozyme | Placebo
Number analyzed (Participants) | 5 | 6
units on a scale | 5.875 [-0.436 to 12.19] | 3 [0.055 to 5.945]
Statistical Analysis 1: Comparison: Pulmozyme vs Placebo; Test type: Superiority or Other; p = 0.2, t-test, 2 sided — P-value of < 0.05 is considered significant

2. Primary Outcome: Improvement in Appearance of Nasal Passages/Sinuses
Description: periodic endoscopic photos of sinuses by ear-nose-throat (ENT) surgeon. The scale for scoring severity of disease ranges from 0 (best possible outcome) to 2 (worst possible outcome).
  independent blinded scoring by 2 surgeons difference in scores pre and post are reported (1 year minus baseline)
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: units
Groups:
- Pulmozyme: endoscopic photos of sinuses by ENT surgeon independently and blindly scored by two surgeons with scale of 0,1,2 to indicate severity of disease
- Placebo: endoscopic photos of sinuses by ENT surgeon, independently and blindly scored by two surgeons. Scores of 0,1,2 based on disease severity.
Arm/Group | Pulmozyme | Placebo
Number analyzed (Participants) | 5 | 6
units | 0.2 [-0.84 to 1.24] | -1 [-2.24 to 0.24]
Statistical Analysis 1: Comparison: Pulmozyme vs Placebo; Test type: Superiority or Other; p = 0.048, t-test, 2 sided — P-value of < 0.05 is considered significant

3. Secondary Outcome: Chronic Sinusitis Survey Score
Description: pre-surgery and end of trial (12 months) Reduction in scores (baseline minus 1 year) are recorded The chronic sinusitis survey consists of 6 questions, ranges from 0-24, a lower score indicates the best possible outcome.
Time Frame: baseline and 1 year
Measure: Mean (95% Confidence Interval); unit: units on a scale
Groups:
- Pulmozyme: Scores from the Chronic Sinusitis Survey
- Placebo: Scores from the Chronic Sinusitis Survey recorded
Arm/Group | Pulmozyme | Placebo
Number analyzed (Participants) | 5 | 6
units on a scale | 8.5 [5.45 to 11.55] | 3 [-1.92 to 7.92]
Statistical Analysis 1: Comparison: Pulmozyme vs Placebo; Test type: Superiority or Other; p = 0.003, t-test, 2 sided — P-value < 0.05 is considered significant

4. Secondary Outcome: Pulmonary Function
Description: prior to surgery and end of study spirometry as measured by forced expiratory volume in 1 second (FEV1) percent predicted. The change over the course of the study (1 year minus baseline) is reported. A higher value indicates a better outcome.
Time Frame: baseline and 1 year
Measure: Mean (Full Range); unit: percentage of predicted FEV1
Groups:
- Pulmozyme: Percent predicted for forced expiratory volume in 1 second recorded
- Placebo: Percent predicted forced expiratory volume in 1 second recorded
Arm/Group | Pulmozyme | Placebo
Number analyzed (Participants) | 5 | 6
percentage of predicted FEV1 | 0.8 [-20 to 17] | 5.4 [-3 to 18]
Statistical Analysis 1: Comparison: Pulmozyme vs Placebo; Test type: Superiority or Other; p = 0.4, t-test, 2 sided — P <0.05 is considered significant

ADVERSE EVENTS:
Time Frame: 1 year (study period)
Groups:
- Pulmozyme: patients receiving once daily intranasal Pulmozyme
- Placebo: patients receiving once daily intranasal placebo
Arm/Group | Pulmozyme | Placebo
Serious Adverse Events (participants affected / at risk) | 1/8 | 2/8
Other Adverse Events (participants affected / at risk) | 1/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmozyme (N=8) | Placebo (N=8)
hospitalization for pulmonary exacerbation (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pulmozyme (N=8) | Placebo (N=8)
sinus surgery (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
recruitment for a long trial was difficult so enrollment was truncated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less